CLINICAL TRIAL: NCT06582875
Title: Advancing ADPKD Treatment With GLP-1RA: A Study of Glucagon-Like Peptide-1 Receptor Agonists' Efficacy, Safety, and Mechanism
Brief Title: Glucagon-Like Peptide-1 Receptor Agonist in ADPKD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Washington University School of Medicine (Other); Mayo Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-0594; R01DK138915-01A1 (NIH)
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Autosomal Dominant Polycystic Kidney; Obesity
Keywords: GLP1RA
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): To minimize the risk of gastrointestinal adverse events, we will use a standard dose-escalation regimen for tirzepatide (placebo-matched), starting at 2.5 mg once weekly (OW) at randomization. After 4 weeks of treatment at 2.5 mg, the dose will be escalated to 5 mg OW, which will be maintained for another 4 weeks and then continued as the target dose for 10 months until the end of treatment. As with other nutrient stimulating hormone (NuSH) therapies, dose reductions and extensions of dose-escalation intervals will be permitted if participants experience unacceptable adverse events. The minimum tolerated dose required for continued study participation is 2.5 mg/week. All dose changes will be documented in the study records.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): To minimize the risk of gastrointestinal adverse events, we will use a standard dose-escalation regimen for tirzepatide (placebo-matched), starting at 2.5 mg once weekly (OW) at randomization. After 4 weeks of treatment at 2.5 mg, the dose will be escalated to 5 mg OW, which will be maintained for another 4 weeks and then continued as the target dose for 10 months until the end of treatment. As with other nutrient stimulating hormone (NuSH) therapies, dose reductions and extensions of dose-escalation intervals will be permitted if participants experience unacceptable adverse events. The minimum tolerated dose required for continued study participation is 2.5 mg/week. All dose changes will be documented in the study records.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Titrated to dose of 5 mg once weekly subcutaneous
  Other Names: Zepbound
  Arms: Tirzepatide
Other: Placebo — Titrated to dose of 5 mg once weekly subcutaneous
  Arms: Placebo

SUMMARY:
The proposed clinical trial aims to assess if a year of treatment with a glucagon-like peptide 1 receptor agonist, a medication approved for weight management that also improves the body's response to glucose and insulin, can slow kidney growth in adults with autosomal dominant polycystic kidney disease who are overweight or obese. The study will also evaluate changes in abdominal fat and kidney metabolism using cutting-edge images techniques. Blood and urine samples will provide further insight into biological changes that may be linked to the benefits of the intervention, while ensuring careful monitoring of safety and tolerability.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is a common inherited disorder that leads to kidney failure. The only approved treatment to decelerate kidney disease progression in patients with ADPKD is tolvaptan, but its usage is limited due to frequent side effects affecting adherence. Thus, alternative interventions that may slow ADPKD progression hold considerable clinical importance. In line with the general population, body-mass index and insulin resistance have been increasing in patients with ADPKD. The investigators have shown that visceral adiposity associates strongly with accelerated progression of early-stage ADPKD. Pilot study suggested that diet-induced weight loss may slow kidney growth (% in height-adjusted total kidney volume [htTKV] by magnetic resonance imaging), and the study team is currently evaluating the efficacy of daily caloric restriction-induced weight loss for slowing ADPKD progression in a phase IIa clinical trial. However, the long-term adherence to lifestyle interventions is challenging, making pharmacological interventions a compelling adjunct or alternative. Moreover, the study team recently demonstrated that adults with ADPKD and preserved kidney function exhibited insulin resistance (via the gold-standard hyperinsulinemic-euglycemic clamps) and impaired kidney oxidative metabolism (via 11C-acetate PET), which were strongly associated with htTKV. These novel data suggest that targeting improvements in insulin sensitivity and kidney oxidative metabolism, in addition to weight loss, may slow ADPKD progression. Glucagon-like peptide 1 receptor agonists (GLP-1RAs) were recently FDA-approved for the treatment of obesity and show promise in substantially reducing adiposity and improving insulin sensitivity. Additionally, evidence indicates that GLP-1RAs may transform CKD management by reducing kidney events in patients with and without diabetes, via effects extending beyond glycemic modulation, and in part via attenuated kidney inflammation and oxidative stress. However, GLP-1RAs have not yet been evaluated as a novel therapy for slowing ADPKD progression in patients with overweight/obesity. Thus, the current study is a 12-month, phase II, randomized, placebo-controlled, double-blind clinical trial using a GLP-1RA in 126 adults with ADPKD and overweight or obesity to slow kidney growth (primary outcome). The trial will also evaluate changes in total body weight, adipose volume and function, insulin resistance, kidney oxidative metabolism, and inflammation, and carefully monitor safety and tolerability. As a novel therapeutic in ADPKD, GLP-1RAs could transform the treatment landscape for patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* ADPKD diagnosis based on the modified Pei-Ravine criteria
* Body-mass index of ≥27 kg/m^2
* Estimated glomerular filtration rate ≥ 30 mL/min/1.73m^2
* Mayo Classification of C, D, or E, calculated from a previous kidney ultrasound or MRI performed within the last 12 months
* Not currently participating in or planning to participate in any formal weight loss or physical activity program, or another interventional study
* Ability to provide informed consent

Exclusion Criteria:

* Diabetes mellitus
* Tolvaptan usage or plans to initiate tolvaptan
* History of hospitalization or major surgery within the last 3 months
* Uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure >100 mm Hg)
* Pregnancy, lactation, or unwillingness to use adequate birth control
* Regular use of prescription or over-the-counter medications that may affect weight, appetite, food intake, or energy metabolism
* History of clinically diagnosed eating disorder including: anorexia nervosa, bulimia, binge eating disorder
* Weight change of >5% in the past 3 months for any reason except post-partum weight loss
* Inability to cooperate with or clinical contraindication for MRI including: severe claustrophobia, implants, devices, or non-removable body piercings
* Presence or personal history of malignant neoplasm within 5 years prior to the day of screening
* Personal or family history of medullary thyroid carcinoma, thyroid nodule, or multiple endocrine neoplasia type 2
* Prior history of pancreatitis
* Weight ≥450 lb

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in height-Adjusted Total kidney volume | Baseline, 12-months
  To assess kidney growth,height-adjusted total kidney volume will be measured by magnetic resonance imaging at baseline and 12 months to determine annual percent change.

SECONDARY OUTCOMES:
Change in body weight | Baseline, 12-months
  Change in body weight over the 12-month period will be measured using a calibrated digital scale.
Change in abdominal adiposity | Baseline, 12-months
  Abdominal adiposity (subcutaneous, visceral, and total) will be assessed by magnetic resonance imaging.
Change in adiponectin (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in leptin (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in interleukin-6 (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in tumor necrosis-factor-alpha (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in high-sensitivity C-reactive protein (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in 8-isoprostane (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in copeptin (circulating) | Baseline, 6-months, 12-months
  Venous blood samples will be analyzed for this mechanistic biomarker
Change in HOMA-IR | Baseline, 6-months, 12-months
  The Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will use fasting glucose and insulin to calcuate insulin sensitivity
Change in HOMA-β | Baseline, 6-months, 12-months
  The Homeostatic Model Assessment of β-cell function (HOMA-β) will use fasting glucose and insulin to calcuate insulin secretion.
Change in 8-isoprostane (urinary) | Baseline, 6-months, 12-months
  Sport urine samples will be analyzed for this mechanistic biomarker
Change in copeptin (urinary) | Baseline, 6-months, 12-months
  Sport urine samples will be analyzed for this mechanistic biomarker
Change in renal oxygen consumption | Baseline, 12-months
  Renal oxygen consumption will be assessed by a PET/CT scan using 11-C acetate in a sub-set of participants
Change in gut microbiota | Baseline, 12-months
  16S rRNA gene sequencing will be used for taxonomic characterization of the gut microbiota in a subset of participants.

OTHER OUTCOMES:
Change in renal blood flow | Baseline, 12-months
  Phase contrast magentic resonance imaging will be used to measure change in renal blood flow
Safety (adverse events) | 12 months
  Number of participants with treatment-related adverse events in each group as evaluated by the DSMB
Adherence | 12 months
  Compliance will be assessed by cross-checking the following sources and comparing these to the expected use: (1) drug accountability information; (2) counting returned trial product, visual inspection of pens; and (3) discussion with participants.
Tolerability (dropout due to adverse events) | 12 months
  Subject dropout due to treatment-emergent adverse events
Kidney Function Decline | Baseline, 1 month, 3 months, 6-months, 12-months
  Estimated glomerular filtration rate trajectories will be compared between the active and placebo group as an exploratory endpoint to inform a subsequent phase III trial.
Change in dietary energy Intake | Baseline, 1 month, 6-months, 12-months
  Multiple pass 24-hr dietary recalls will be analyzed to evaluate self-reported energy intake
Change in free-living physical activity | Baseline, 12-months
  Estimated energy expenditure (METs) over a 7-day period will be quantified using the ActiGraph wGT3X-BT activity monitor
Change in resting energy experniture | Baseline, 12 months
  Resting energy expenditure will be assessed using indirect calorimetry.
Change in percent body fat | Baseline, 12 months
  Percent body fat will be assessed via DEXA scan in a sub-set of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in ADPKD. Data shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. data use agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Derived] Cortinovis M, Perico N, Remuzzi G. The Need for Novel Therapeutic Directions in Autosomal Dominant Polycystic Kidney Disease Patient Care. Clin J Am Soc Nephrol. 2025 Dec 5. doi: 10.2215/CJN.0000000975. Online ahead of print. PMID 41348481